CLINICAL TRIAL: NCT06915714
Title: The Prognostic Value of Quantitative Parameters Derived From Dual Scanning of FDG and PSMA PET/CT for Tumor Progression in Patients With Metastatic Hormone-sensitive Prostate Cancer Receiving Novel Hormone Therapy
Brief Title: The Prognostic Value of PET/CT for Tumor Progression in Patients With Metastatic Hormone-sensitive Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zheng fufu, Professor, Phd, Md, Sun Yat-sen University
Other Study IDs: IIT-2025-117
Record Dates: First submitted 2025-03-22; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer Metastatic Disease; PET / CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group1: PCa40%MTV-P = High, PCa40%MTV-G = Low
- Group2: PCa40%MTV-P = Low, PCa40%MTV-G = High
- Group3: PCa40%MTV-P = Low, PCa40%MTV-G = Low
- Group4: PCa40%MTV-P = High, PCa40%MTV-G = High

SUMMARY:
Investigators retrospectively collected data from consecutive patients treated at the First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China, from October 2020 to March 2024. The inclusion criteria were as follows: (1) patients with diagnosis of metastatic hormone-sensitive prostate cancer, confirmed by PSA levels, radiographic tests and pathological information; (2) patients who underwent FDG and PSMA PET/CT prior to the initiation of medical treatment. The exclusion criteria were as follows: (1) patients who received novel hormone therapy or a prostate biopsy prior to PET/CT; (2) patients with other malignancies; (3) patients received hormone therapy without NHT; (4) patients received chemotherapy or radiotherapy prior to or during novel hormone therapy; (5) absence of follow-up data at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of metastatic hormone-sensitive prostate cancer, confirmed by PSA levels, radiographic tests and pathological information
* patients who underwent FDG and PSMA PET/CT prior to the initiation of medical treatment

Exclusion Criteria:

* patients who received novel hormone therapy or a prostate biopsy prior to PET/CT
* patients with other malignancies
* patients received hormone therapy without novel hormone therapy
* patients received chemotherapy or radiotherapy prior to or during novel hormone therapy
* absence of follow-up data at our institution

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the enrolled patients were Asian(we are a affiliated hospital of a university based in Mainland china ).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-06-02 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Castration-Resistant Prostate Cancer free survival (CRPC-FS) | From date of the initiation of novel hormone therapy until the date of first documented either PSA or radiography-confirmed progression or date of the last follow-up for any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Fangzheng Xiang, Principal Investigator — First affiliated hospital, Sun Yat-sen univeristy
Locations (1):
- First affiliated hospital, Sun Yat-sen univeristy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No